CLINICAL TRIAL: NCT02121041
Title: Comparative Effectiveness of Ambulatory Blood Pressure Monitoring vs Usual Care for Diagnosing and Managing Hypertension: A Pilot Study
Brief Title: Ambulatory vs Office BP Management Usual Care for Diagnosing and Managing Hypertension: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anthony J Viera, MD, MPH (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor-Investigator, Anthony J Viera, MD, MPH, Distinguished Associate Professor, Family Medicine, University of North Carolina, Chapel Hill
Organization: University of North Carolina, Chapel Hill (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 14-0670
Record Dates: First submitted 2014-04-16; First posted 2014-04-23 (Estimated); Results first posted 2016-12-19 (Estimated); Last update posted 2017-02-10 (Actual); Status verified 2016-12

CONDITIONS: Hypertension
Keywords: Hypertension; Blood Pressure; Ambulatory Blood Pressure Monitoring
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Chlorthalidone; Losartan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual Care (No Intervention): Participants in the usual care arm will have 2 ABPM sessions during the study, but ABPM will not be used to make a diagnosis or dictate anti-hypertensive treatment. Any recommendations for anti-hypertensive treatment will be made only via regular clinical care.
- ABPM Guided (Active Comparator): Participants in the ABPM-guided arm will undergo 3 ABPM sessions. Results of ABPM will be used to make diagnoses and dictate anti-hypertensive treatment as applicable. Anti-hypertensive medications may include: Amlodipine, Chlorthalidone and/or Losartan.
  Interventions: Drug: Amlodipine; Drug: Chlorthalidone; Drug: Losartan

INTERVENTIONS:
Drug: Amlodipine — Amlodipine 5 mg or 10 mg
  Other Names: Norvasc
  Arms: ABPM Guided
Drug: Chlorthalidone — Chlorthalidone 12.5 mg or 25 mg
  Other Names: Thalitone
  Arms: ABPM Guided
Drug: Losartan — Losartan 50 mg or 100 mg
  Other Names: Cozaar
  Arms: ABPM Guided

SUMMARY:
The purpose of this study is to compare the effectiveness of ambulatory blood pressure monitoring to usual care (blood pressure measurement in the office) in diagnosing and managing hypertension.

DETAILED DESCRIPTION:
The usual strategy for detecting hypertension-repeated office blood pressure (BP) measurements-is inefficient and inaccurate. When paired with ambulatory BP monitoring (ABPM), which takes a multitude of measurements over 24 hours, it is clear that office BP measurements may convey a falsely positive diagnosis known as white-coat hypertension. What is less well-known is that office BP measurements may also convey a falsely negative diagnosis termed masked hypertension (MH). That is, office BP may measure as normal, yet 24-hour ambulatory measurements show elevated BP. People with MH have cardiovascular risk that is similar to that of people with diagnosed hypertension, yet MH goes unrecognized, and therefore, untreated. Ultimately, identifying the best strategy for accurately detecting hypertension is vital to improving overall BP control and reducing cardiovascular events. Without a feasible ABPM strategy, MH will continue to go unrecognized and untreated.

Participants enrolled in the study will be randomized to either the usual care group or the ABPM-guided group. All participants will have a baseline ABPM. ABPM will be used to make a diagnosis and determine anti-hypertensive treatment in the ABPM-guided group only. Participants in the ABPM-guided group will have a follow-up ABPM in 2 months. All participants will have a final ABPM 4 months after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 30 years and ≤ 65 years
* Most recent (within 14 days) clinic systolic BP 126-150 mm Hg
* Able/willing to wear a BP monitor for 24 hours on multiple occasions
* Able/willing to take daily anti-hypertensive medication if indicated
* Able to read and speak English

Exclusion Criteria:

* Pregnant or trying to become pregnant
* Known heart disease
* History of persistent atrial fibrillation
* Currently taking antihypertensive medication
* Currently taking Simvastatin > 20mg daily
* Clinician recommends against participation

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2014-05; Primary Completion 2015-09 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Viera, MD, MPH, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care | ABPM Guided
Started | 14 | 14
Completed | 13 | 8
Not Completed | 1 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care | ABPM Guided | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Customized [Mean (Standard Deviation); unit: years] | 47.6 (12) | 49.2 (10) | 48.4 (11)
Gender [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 6 | 7 | 13

OUTCOME MEASURES:

1. Primary Outcome: 24 Hour Blood Pressure Average at the End of 4 Month Participation.
Time Frame: Participants will be on study average of 4 months.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Usual Care | ABPM Guided
Number analyzed (Participants) | 13 | 8
mm Hg | 134 (11) | 132 (10)

ADVERSE EVENTS:
Arm/Group | Usual Care | ABPM Guided
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14
Other Adverse Events (participants affected / at risk) | 1/14 | 1/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Usual Care (N=14) | ABPM Guided (N=14)
electrolyte (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — Abnormal electrolyte level

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No